CLINICAL TRIAL: NCT03902782
Title: Ultrasound-Guided Erector Spinae Plane Block Versus Intercostal Nerve Block For Postoperative Pain Control in Video-Assisted Thoracoscopic Surgery: A Prospective, Double Blind Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Intercostal for VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor of anesthetsia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-5553
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases | interventions — Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block (Experimental): patients will receive an ultrasound guided ESP block (technique as described by Forero et al) under strict sterile conditions in the operating room area. After identifying the T5 transverse process (TP) and after infiltration of lidocaine 2% subcutaneously. A 22g 100mm block needle will be advanced under vision, in a cephalad to caudad direction, until the tip contacts the T5 TP. 20 ml of 0.25% bupivacaine with 5 mcg/ml of epinephrine and 10 mg dexamethasone will be injected under the erector spinae muscle. A visible separation of the erector spinae muscle from the TP will be the sign of a successful block. A 20 ml syringe of Normal Saline will be given to the surgeon (unaware of the content) at the end of the surgery, for the intercostal nerve block as per standard present technique.
  Interventions: Procedure: ESP block; Procedure: Sham Intercostal block; Drug: Bupivacaine-epinephrine; Drug: Dexamethasone injection; Drug: Normal saline
- ESP sham block (Sham Comparator): patients will receive an ultrasound guided sham ESP block under strict sterile conditions in the operating room area as described above. 20 ml of Normal Saline will be injected under the erector spinae muscle. A 20 ml syringe of 0.25% bupivacaine with 5 mcg/ml of epinephrine and 10 mg dexamethasone will be given to the surgeon (blinded to the content) at the end of the surgery for the intercostal nerve block.
  Interventions: Procedure: Intercostal block; Procedure: Sham ESP block; Drug: Bupivacaine-epinephrine; Drug: Dexamethasone injection; Drug: Normal saline

INTERVENTIONS:
Procedure: ESP block — ESP with 20 ml of Bupivacaine 0.25%, Epinephrine 5mcg/ml and Dexamethasone 10mg.
  Sham intercostal block with 20 ml Normal Saline
  Arms: ESP block
Procedure: Intercostal block — Intercostal block with 20 ml of Bupivacaine 0.25%, Epinephrine 5mcg/ml and Dexamethasone 10mg.
  Sham ESP with 20 ml Normal Saline
  Arms: ESP sham block
Procedure: Sham ESP block — As described earlier
  Arms: ESP sham block
Procedure: Sham Intercostal block — As described earlier
  Arms: ESP block
Drug: Bupivacaine-epinephrine — As described earlier
Drug: Dexamethasone injection — As described earlier
Drug: Normal saline — As described earlier

SUMMARY:
The Erector Spinae Plane (ESP) block is a new interfascial regional anesthesia technique recently described by Forero et al. Currently the literature shows the ESP block being used for analgesia after thoracic surgery, breast surgery, abdominal surgery (visceral abdominal analgesia in bariatric surgery, ventral hernia repair, cholecystectomy), thoracic vertebral surgery and for pain relief in rib fractures. Taking in consideration the excellent clinical experience, but the lack of strong and high-quality evidence, supporting the use of ESP block for pain management in patients undergoing VATS procedures, there is a specific interest to develop a prospective study. Comparing the effect of the current pain relief strategy at the MGH (intercostal nerve block by the surgeon at the end of the procedure ) versus ESP block after VATS, seems warranted to improve current clinical results.

DETAILED DESCRIPTION:
In recent years, Video-Assisted Thoracic surgeries (VATS) has become the preferred approach for thoracic surgeries over thoracotomies, due to its clear advantages, such as improved pulmonary function, rapid recovery and reduced pain scores postoperatively. Although pain is reduced in VATS when compared to conventional thoracotomies, patients still experience moderate to severe pain, mainly due to intercostal nerve damage by ports and drains, as well as the surgical resection itself. Adequate pain relief leads to earlier and better mobilization, improves respiratory functions, and decreases global stress response. In addition, it helps in reducing the chances of developing chronic postoperative pain.

Epidural blockade has been recognized as the gold standard for analgesia in thoracic surgeries, with paravertebral blocks (PVB) replacing that standard in VATS procedures, due it's less deleterious adverse effects. Nevertheless, paravertebral blockade still poses some adverse effects such as pneumothorax and the risk of an epidural blockade. Moreover, it might prove difficult to perform in the untrained hand. Thus, a simpler blockade is warranted in patients undergoing VATS.

Proper pain relief is critical in the early postoperative period in VATS surgery, to allow early discharge of patients according to the clinical pathway milestones. The excessive consumption of opioids to achieve this goal on the other hand, may produce complications and side effects not compatible with the early discharge plan.

The Erector Spinae Plane (ESP) block is a new interfascial regional anesthesia technique recently described by Forero et al . It consists of injecting 20 ml of local anesthetic (ie.: ropivacaine 0.5%), under ultrasound guidance, at the level of the T5 transverse process in the tissue plane deep to the erector spinae muscle. A study on the ESP block was conducted on fresh human cadavers; dye mixture was injected deep to erector spinae muscle, and the spread showed to be cranio-caudal from C7 to T8, lateral spread extended to the tips of the transverse processes at all levels, penetration of the dye was beyond the costotransverse junction and anteriorly into the inter transverse spaces. In addition, there was evidence of dye penetration deep to the intercostal muscles and into the immediate vicinity of the ventral and dorsal rami of the spinal nerve roots. The authors discussed the most significant advantage of the ESP block is its simplicity and safety. The sonoanatomy is easily recognizable, there are no structures at risk of needle injury in the immediate surroundings (lower risk of nerve damage and pneumothorax), and is probably safer for patients with coagulation disorders. The technique also allows the insertion of an indwelling catheter to extend the duration of analgesia as needed.

Currently the literature shows the ESP block being used for analgesia after thoracic surgery, breast surgery, abdominal surgery (visceral abdominal analgesia in bariatric surgery, ventral hernia repair, cholecystectomy), thoracic vertebral surgery and for pain relief in rib fractures.

Taking in consideration the excellent clinical experience, but the lack of strong and high-quality evidence, supporting the use of ESP block for pain management in patients undergoing VATS procedures, there is a specific interest to develop a prospective study. Comparing the effect of the current pain relief strategy at the MGH (intercostal nerve block by the surgeon at the end of the procedure ) versus ESP block after VATS, seems warranted to improve current clinical results.

In this randomized controlled trial, the investigator hypothesize that a single injection ESP block, would provide an effective post operative pain relief, superior to an intercostal nerve block, in patients undergoing VATS procedures.

The study will be conducted at the Montreal General Hospital, one hundred patients; ASA I-III male and female patients aged between 18 to 80 years old, who are scheduled for Video assisted thoracic surgery. Patients will be recruited before surgery. Informed consent will be obtained by a Research Assistant.

Patients will be prospectively randomized in a double blind fashion, using a computer-generated number placed in a sealed brown envelope, into either group 1, receiving ESP block, or group 2, receiving sham ESP block.

In group 1, patients will receive an ultrasound guided ESP block (technique as described by Forero et al) under strict sterile conditions in the operating room area. After identifying the T5 transverse process (TP) and after infiltration of lidocaine 2% subcutaneously. A 22g 100mm block needle will be advanced under vision, in a cephalad to caudad direction, until the tip contacts the T5 TP. 20 ml of 0.25% bupivacaine with 5 mcg/ml of epinephrine and 10 mg dexamethasone will be injected under the erector spinae muscle. A visible separation of the erector spinae muscle from the TP will be the sign of a successful block. A 20 ml syringe of Normal Saline will be given to the surgeon (unaware of the content) at the end of the surgery, for the intercostal nerve block as per standard present technique.

In group 2, patients will receive an ultrasound guided sham ESP block under strict sterile conditions in the operating room area as described above. 20 ml of Normal Saline will be injected under the erector spinae muscle. A 20 ml syringe of 0.25% bupivacaine with 5mcg/ml of epinephrine and 10 mg dexamethasone will be given to the surgeon (blinded to the content) at the end of the surgery for the intercostal nerve block.

All medications will be prepared by a research assistant not assigned to the case, and not involved in the follow up assessment. Two 20 ml syringes will be prepared under sterile precautions, one containing Bupivacaine 0.25% with epinephrine 5 µg/ml and 10 mg dexamethasone, and the other containing 0.9% normal saline. Syringes will be labeled as "ESP" and "intercostal" according to the randomization. The evaluator in the postoperative period, the anesthesiologist, the patient and the surgeon will be blinded to the group randomization.

General anesthesia will be induced with propofol 1.5-2 mg/kg and fentanyl 2 mcg/kg, as well as rocuronium 0.6 mg/kg to facilitate tracheal intubation with a double lumen tube (DLT). A 3.2 mm fiberoptic bronchoscope will be used to confirm correct placement of the DLT, to allow one lung ventilation intraoperatively. Anesthesia will be maintained with sevofluorane or desflourane according to the anesthesiologist's preference.

For intra-operative analgesic requirements, Specific instructions will be handed to each anesthetist to administer fentanyl 25 mcg increments every 5 minutes in the following scenarios:

Elevation in the heart rate of more than 20% of baseline values. Elevation in blood pressure of more than 20% of baseline values.

Patients will receive Ondansetron 4mg prior to extubation. Post anesthetic care and medications will include.

Acetaminophen 975mg, PO or PR, Q6H Celecoxib 100mg, PO, BID for 5 days Ondansetron 4mg, PO or IV, Q8H, PRN (for nausea or vomiting) Nalbuphine 2.5 mg, IV, diluted PRN (for pruritus) Polyethylene glycol 17gr, PO, Day, PRN (for constipation)

All patients enrolled will be provided with a Patient Controlled Analgesia (PCA) pump for first 24 hours after the surgery. The pump will be programmed to deliver Morphine sulfate 1mg, lockout time 7 min, without a continuous infusion rate, capable to be increased to 1.5mg if pain VAS≥7 with the absence of sign or symptoms of toxicity. Hydromorphone will be used in case of Morphine allergy. Patients will be clearly instructed to trigger the PCA Only if they perceive pain as >4/10 If the PCA IV line gets lost with failure to obtain a new one, in patients with VSA>4, a rescue dose 3-5mg morphine SC Q4H PRN will be considered. The time and dose of rescue medication will be recorded.

The Standard Institutional Postoperative Clinical Pathway will be followed in both groups, except for the use of PCA.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* age between 18 to 80 years old
* ASA 1-3
* scheduled for VATS
* informed consent explained and signed

Exclusion Criteria:

* Patients < 18 years old, > 80 years old
* ASA physical status > 3
* morbid obesity (BMI >40)
* previous cardiac surgery or ipsilateral thoracic surgery
* neuropsychiatric diseases
* serum albumin < 35 g/L
* cardiac, renal (creatinine > 200mmol/l) or hepatic failure (aspartate amino transferase, alanine amino transferase > 50 % over the normal range)
* anemia (hematocrit <30%)
* organ transplant
* allergy to analgesics or local anesthetics or other medications used in the study
* abuse of opioids or sedatives
* contraindication to receive regional anesthesia (e.g. coagulation defect)
* patients who could not understand the VAS pain-scoring system
* patient refusal to follow participation
* intraoperative conversion to open thoracotomy
* revision or re-operation or complication of surgery during the follow-up time
* post operative mechanical ventilation
* intolerance or allergy to any prescribed medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of ESP block versus Intercostal nerve block in decreasing opioid consumption | Measured at 24 hours postopertively
  measured by total intravenous morphine consumption at 24 hours postopertively. A 25% reduction in morphine consumption would be considered statistically significant.

SECONDARY OUTCOMES:
Efficacy of ESP block versus Intercostal nerve block in decreasing pain intensity at rest: Numerical Rating Scale (NRS) | measured at post operative 2, 4, 12, 24 and 48 hours
  Pain levels will be assessed using the 10 points Numerical Rating Scale (NRS) where zero= no pain and 10= pain as bad as it can be. The NRS is a validated tool to measure pain and discomfort. It is sensitive to pharmacological and non-pharmacological interventions, that have an impact over the experience of pain, as well as it's high correlation with pain levels
Efficacy of ESP block versus Intercostal nerve block in decreasing pain intensity upon mobilization: Numerical Rating Scale (NRS) | measured at post operative 2, 4,12, 24 and 48 hours
  Pain levels will be assessed using the 10 points Numerical Rating Scale (NRS) where zero= no pain and 10= pain as bad as it can be. The NRS is a validated tool to measure pain and discomfort. It is sensitive to pharmacological and non-pharmacological interventions, that have an impact over the experience of pain, as well as it's high correlation with pain levels
Change in pulmonary function | pre-operatively and 2, 4, 12, 24 and 48 hours after the procedure
  This will be assessed using the incentive spirometer, which allows for crude measurement of inspired volumes
Total opioid consumption | 48 hours post operatively
  In morphine equivalencies
Ipsilateral shoulder pain scores | 2, 4, 12, 24 and 48 hours after the procedure
  Pain levels will be assessed using the 10 points Numerical Rating Scale (NRS) where zero= no pain and 10= pain as bad as it can be. The NRS is a validated tool to measure pain and discomfort. It is sensitive to pharmacological and non-pharmacological interventions, that have an impact over the experience of pain, as well as it's high correlation with pain levels
Incidence of adverse events | Over the first 48 hours
  postoperative nausea and vomiting (PONV), hypotension, urinary retention (requiring placement of an indwelling or a temporary catheter), pruritis and oxygen requirements
Length of stay in the post anesthesia care unit (PACU) | up to 24 hours
  total time spent in the PACU until reaching PACU discharge criteria
Length of stay in the hospital | up to 10 days
  total time spent in the hospital until reaching hospital discharge criteria
Time to first mobilization to the chair | Measured from the arrival time to PACU
Time to first ambulation (walking) out of bed | Measured from the arrival time to PACU
Block performance time | Up to 40 minutes
  The time it takes to perform the ESP block
Block related adverse events | First 4 hours postopertively
  Incidence of block related adverse events such as bleeding, pneumothorax and local anesthetic systemic toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided